CLINICAL TRIAL: NCT05459493
Title: The Efficacy and Safety of Chinese Herbal Compound TJAOA101 in Treatment of Diminished Ovarian Reserve: a Prospective, Multi-center and Before-after Study.
Brief Title: A Clinical Study of Chinese Herbal Compound TJAOA101 in Therapy of Diminished Ovarian Reserve
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Shixuan Wang, Professor, Tongji Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TJ-IRB20220634-DOR
Record Dates: First submitted 2022-06-29; First posted 2022-07-15 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Diminished Ovarian Reserve
Keywords: Diminished Ovarian Reserve; Traditional Chinise Medicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TJAOA101 (Experimental): Once enrolled, participants will be administrated TJAOA101 and followed by a 3-month medication cycle. The usage of this herbal compound is to take orally twice a day(two sacks per). Add it to about 200ml warm water and take it half an hour before breakfast in the morning and half an hour before bedtime in the evening except menstrual period.
  Interventions: Drug: TJAOA101

INTERVENTIONS:
Drug: TJAOA101 — Once enrolled, participants will be administrated TJAOA101

SUMMARY:
Currently, no drugs have been developed for DOR. We developed the Chinese herbal compound TJAOA101 and has validated its effects in animals. Here, we will perform a population-based, multicenter study to confirm the safety and efficacy of TJAOA101 in therapy of DOR. We aim to provide a solid evidence for TCM in therapy of DOR.

DETAILED DESCRIPTION:
As the pivotal reproductive organ, the ovaries have two main functions: ovulation and secretion of hormones. Ovarian dysfunction not only cause reproductive detriment, but also harms to each system and organ, arousing extensive concern of women. Diminished ovarian reserve (DOR) refers to the decline in ovarian function in advance with reduction of functional follicles and the ability to produce high quality oocytes, resulting in reduced fertility and the lack of sex hormones, leading to early menopause and infertility, and accelerated multiple organ aging including osteoporosis, cardiovascular disease, cognitive impairment. As DOR is an early stage of ovarian dysfunction, early intervention is necessary.

Currently, several therapeutic approaches could be considered to prevent and attenuate unfavorable consequences of ovarian function decline. The hormone replacement therapy (HRT) can add exogenous sex hormones by replenishing the lack of hormones to relieve the symptoms caused by low level of estrogen, and then improve the health and life quality. HRT may can bring some benefits to women with DOR. However, it also has some limitations, for instance, it is mainly used for alleviating menopausal symptoms, while not to improve ovarian function. And there are some contraindications, such as breast cancer and blood clots, and HRT may increase the risk of abnormal uterine bleeding(AUB). In addition, dehydroepiandrosterone (DHEA), growth hormone(GH) and aspirin are considered the alternative treatments of DOR. However, due to the lack of large randomized controlled trials, the effectiveness of them needs further confirmation.

Traditional Chinese medicine (TCM) has its own characteristic and superiority in treating diseases, with light side effects and remarkable curative effect. The Chinese nation accumulated a great deal of experience in TCM for treating ovarian dysfunction. Several studies showed that TCM is effective and safe in treating DOR. However, no guidelines for long-term TCM management in treating ovarian function decline exist at present. Clinical trials are imperative to test the safety and efficacy of these TCM prescriptions. And many prescriptions are complicated, mainly rely on the old experience with lacking sufficient scientific basis.

To address this question, we have invented a brand new TCM prescription to treat DOR. Previously, we collected clinical TCM prescriptions from literature retrieval (CNKI and PubMed), and then created a database of recipes for treating ovarian function decline. By using Traditional Chinese Medicine Inheritance Support System (TCMISS) , key TCM and TCM combinations in DPTP were extracted to identify the candidate Chinese herbs. On this basis, gynostemma pentaphylla were added, efficacy and safety of which has been verified in drosophila and mice. Then, TJAOA101 (Tongji Anti-ovarian aging 101), a new TCM recipe was preliminarily developed by multiple experts of pharmacy and gynecology. And multiple model organisms including drosophila, mice of natural aging and chemotherapy damage were further used to verify the safety and effectiveness of TJAOA101 on ovarian function. Finally, the pharmacological action, dose, synergistic effect and incompatibility were determined.

This study is a multicenter and prospective trial aiming to determine the safety and efficacy of TJAOA101 for preventing among women who were diagnosed with DOR. and aims to provide new strategies for improving ovarian reserve and function for DOR patients by evaluating the safety and efficacy of TJAOA1.

ELIGIBILITY:
Inclusion Criteria:

1. The age range of patient is 18-40 years old.
2. Women with DOR, and wish to improve ovarian function or menopausal syndrome. The diagnostic criteria for DOR is as follows: If two of the following three tests of ovarian reserve function are met, DOR can be diagnosed: bilateral AFC<6; AMH < 1.1 ng/ml; 10 mIU/ml <bFSH<25 mIU/ml.
3. Sign the informed consent form.

Exclusion Criteria:

1. Patient is known to be allergic or unsuitable for the Chinese herbal compound.
2. Women who are pregnant and lactating.
3. Patients had been menopause for more than 1 year.
4. Abnormal uterine bleeding, except ovulation disorders.
5. Women is taking hormone drugs and has stopped taking them within 3 months;
6. Women with endometriosis, myadenosis, submucosal fibroids or the size of non-submucosal fibroids is more than 4 cm.
7. The nature of pelvic mass is unknown.
8. Women with polycystic ovary syndrome, hyperprolactinemia, hyperandrogenemia, diabetes, thyroid and adrenal dysfunction and other endocrine diseases affecting ovulation.
9. Patients with serious primary diseases such as cardiovascular, liver, kidney, lung, biliary, hematopoietic system (Hb<90g/L) and malignant tumor, and psychiatric patients.
10. Patients are participating in other clinical trials or have participated in other clinical trials within the last month.
11. Unsuitable for the study evaluated by the investigator.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
recovery rate of ovarian function | 6 months
  As the definition of DOR is based on AMH or bFSH or AFC, the recovery of ovarian function is also based on the recovery of these indicators. In this study, the recovery of ovarian function is defined as serum AMH increased more than 50%, or serum bFSH decreased more than 50%, or antral follicle count(AFC) increased more than 50% compared with that before treatment，or recover to normal level.

SECONDARY OUTCOMES:
recovery rate of menstruation | 6 months
  two consecutive periods return to normal.

CONTACTS AND LOCATIONS:
Overall Officials: Shixuan Wang, Professor, Study Chair — Department of Obstetrics and Gynecology, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, China